CLINICAL TRIAL: NCT07086443
Title: A Multicenter, Prospective, Randomized Controlled Modified Platform Trial Evaluating Placental Derived Allografts and Standard of Care in the Treatment of Nonhealing Diabetic Foot Ulcers Using Matched Controls
Brief Title: Randomized Evaluation of Nonhealing Diabetic Foot Ulcers With Exclusive Wound Therapy
Acronym: RENEW
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sequence LifeScience, Inc. (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RENEW
Record Dates: First submitted 2025-07-11; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot Ulcer; DFU; Diabetic Foot Ulcer (DFU); Foot Ulcer Due to Type 1 Diabetes Mellitus; Foot Ulcer Due to Type 2 Diabetes Mellitus; Ulcer; Ulcer Foot
MeSH Terms: conditions — Diabetic Foot; Ulcer; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: This study is a multi-center, prospective, matched control clinical study trial evaluating placental derived allografts and standard of care versus standard of care alone in the treatment of nonhealing diabetic foot ulcers. The target ulcers are evaluated weekly by the investigator. The subject is treated once a week, to receive weekly applications of one of seven CAMPs plus SOC for 12 weeks or until the study ulcer has completely closed (i.e. 100% closure as assessed by the investigator and confirmed 2 weeks later at the closure confirmation visit (CCV). One additional visit per week is optional for both arms, for the purpose of changing only the secondary dressing in the CAMP arm. The study utilizes a modified platform design adopted from clinical trials developed during the pandemic to simultaneously test multiple interventions in a single trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Activate™ Matrix +SOC (Experimental): Three layers: amnion, intermediate layer, and chorion
  Interventions: Other: Activate™ Matrix
- AmnioDefend™ FT Matrix +SOC (Experimental): Three layers: amnion, intermediate layer, and chorion
  Interventions: Other: AmnioDefend™ FT Matrix
- Palisade™ DM Matrix +SOC (Experimental): Two layers: amnion and chorion
  Interventions: Other: Palisade™ DM Matrix
- Enclose™ TL Matrix +SOC (Experimental): Three layers: amnion, chorion, amnion
  Interventions: Other: Enclose™ TL Matrix
- Sentry™ SL Matrix +SOC (Experimental): One layer: amnion
  Interventions: Other: Sentry™ SL Matrix
- Shelter™ DM Matrix +SOC (Experimental): Two layers: amnion and chorion
  Interventions: Other: Shelter™ DM Matrix + SOC

INTERVENTIONS:
Other: Activate™ Matrix — Participants will receive weekly applications of Activate™ Matrix and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Activate™ Matrix +SOC
Other: AmnioDefend™ FT Matrix — Participants will receive weekly applications of AmnioDefend™ FT Matrix and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: AmnioDefend™ FT Matrix +SOC
Other: Palisade™ DM Matrix — Participants will receive weekly applications of Palisade™ DM Matrix and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Palisade™ DM Matrix +SOC
Other: Enclose™ TL Matrix — Participants will receive weekly applications of Enclose™ TL Matrix and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Enclose™ TL Matrix +SOC
Other: Sentry™ SL Matrix — Participants will receive weekly applications of Sentry™ SL Matrix and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Sentry™ SL Matrix +SOC
Other: Shelter™ DM Matrix + SOC — Participants will receive weekly applications of Shelter™ DM Matrix and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Shelter™ DM Matrix +SOC

SUMMARY:
The goal of this study is to determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing diabetic foot ulcers with multiple CAMPs plus SOC versus matched controls over 12 weeks using a modified platform trial design.

DETAILED DESCRIPTION:
This study is a prospective modified platform multicenter randomized controlled clinical trial. The goal of this study is to determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing diabetic foot ulcers with multiple CAMPs plus SOC versus matched controls over 12 weeks using a modified platform trial design.

ELIGIBILITY:
Inclusion Criteria:

* The potential subject must be at least 18 years of age or older.
* The potential subject must have a diagnosis of type 1 or 2 Diabetes mellitus.
* At enrollment, the potential subject must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 15.0 cm2 measured post debridement with the imaging device length times width.
* The potential subject must have a target ulcer that has been present for a minimum of 4 weeks of standard of care, prior to the initial screening visit.
* The potential subject must have a target ulcer located on the foot with at least 50% of the ulcer below the malleolus.
* The potential subject must have a target ulcer that is Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
* The potential subject's affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI between 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic. 8. If the potential subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The potential subject must have a target ulcer located on the 50% below the malleolus and not on the dorsal toes.
* The ulcer must be offloaded for at least 14 days prior to enrollment.
* The potential subject must consent to using the prescribed offloading method for the duration of the study.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

* The potential subject is known to have a life expectancy of < 6 months.
* The potential subject's target ulcer is not secondary to diabetes.
* The target ulcer is infected or there is cellulitis in the surrounding skin.
* The target ulcer exposes tendon or bone.
* There is evidence of osteomyelitis complicating the target ulcer.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
* The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
* The surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
* The surface area measurement of the potential subject's target ulcer decreases by 25% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1 visit during which time the potential subject received SOC.
* The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
* The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* The potential subject has participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* The potential subject, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
* The potential subject has a malnutrition.
* The potential subject has a known allergy or sensitivity to PBS, IPA, processing solutions, reagents, or latex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Between-arm difference in subjects achieving complete closure | 1-12 Weeks
  To determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing diabetic foot ulcers with multiple CAMPs plus SOC versus matched controls over 12 weeks using a modified platform trial design.

SECONDARY OUTCOMES:
Time to closure | 1-12 weeks
  To determine the between-arm difference in the time to closure over 12 weeks for CAMP plus SOC versus matched control subjects.
Percentage area reduction rate | 1-12 weeks
  To determine the between-arm difference in percent area reduction (PAR) at weekly intervals for CAMP plus SOC versus matched control subjects.
Adverse Events | 1-12 Weeks
  To determine the between-arm difference in the frequency and nature of adverse events in subjects receiving CAMP plus SOC versus matched control subjects.
Determine quality of life | 1-12 weeks
  To determine the between-arm difference in quality of life for subjects receiving CAMP plus SOC versus matched control subjects using the Forgotten Wound Score (FWS). The FWS is scored on a scale of 0-4. 0 being never and 4 being mostly.
Determine Quality of Life | 1-12 weeks
  To determine the between-arm difference in quality of life for subjects receiving CAMP plus SOC versus matched control subjects Wound Quality of Life (wQOL) questionnaires. WQOL is scored 0-5. 0 being never and 5 being very much.

CONTACTS AND LOCATIONS:
Locations (1):
- Serena Group- Monroeville, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No